CLINICAL TRIAL: NCT02777398
Title: The Prospcetive Randomized Controlled Trial of the Surgical Treatment of Intra-spinal Canal Tumors Using Microsurgical Technique Through Trans-Quadrant Channel Pathway
Brief Title: Surgical Treatment of Intra-spinal Canal Tumors Via Trans-Quadrant Channel
Acronym: STRICT-TAQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-020
Record Dates: First submitted 2016-05-08; First posted 2016-05-19 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Spinal Neoplasms
Keywords: Intra-spinal Canal; Tumor; Minimal Invasive Surgery; Clinical Trial; Quadrant Channel
MeSH Terms: conditions — Spinal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trans-Quadrant Channel Surgery (Experimental): Patients in the experimental arm (experimental group, i.e. microsurgery through trans-Quadrant channel pathway) will be operated using Quadrant channel system. All the tumor resection will be operated through the Quadrant channel with assistance of microsurgical techniques.
  Interventions: Procedure: Trans-Quadrant Channel Surgery
- Conventional Open Surgery (Active Comparator): Patients in the active comparator arm (control group, i.e. conventional open surgery) will be operated using the conventional open surgery. All the tumor resection will be operated directly with conventional procedures. More posterior structures of spine will be removed.
  Interventions: Procedure: Conventional Open Surgery

INTERVENTIONS:
Procedure: Trans-Quadrant Channel Surgery — Patients in the experimental group will be general anaesthetized and placed in the prone position. Intra-operational electrophysiological monitoring will be used. Kirschner wire will be used to identify the position of the Quadrant channel with X-ray. After disinfection and draping, an incision of 3cm long and 2-3cm lateral to midline on the tumor side will be made. Soft tissues will be separated. Graded dilators will be used to establish Quadrant channel. Kerrison clamps will be used to expose the very local posterior spinal structures. Vertebral plate will be windowed with power drill to expose dural mater, and tumors will be removed with microsurgical techniques. Hemostasis will be performed after resection. Dural mater will be closed by titanium clips, and close incision by layers.
  Arms: Trans-Quadrant Channel Surgery
Procedure: Conventional Open Surgery — Patients in the control group will be general anaesthetized during operation and placed in the prone position. Intra-operational electrophysiological monitoring will be used. Surgeons will locate the lesion by X-ray. After disinfection and draping, the midline incision of 7-10 cm and centered by the lesion segment will be made. Soft tissues will be cut and separated to expose posterior structure of spine. The root of spinal process and half of the vertebral plate on tumor side of certain segments will be removed. The dural mater will be opened. Then surgeons will remove tumor with microsurgical techniques. Hemostasis will be precisely performed after resection, and dural mater will be closed by suturing. Incision will be closed by layers. Drainage would be placed if necessary.
  Arms: Conventional Open Surgery

SUMMARY:
Intra-spinal canal tumors are the general term of primary tumors from spinal cord or various tissues in the spinal canal and adjacent to the spinal cord, while the metastatic tumors are those from other sites other than spinal canal. Intra-spinal canal tumor is one of the most common diseases in neurosurgery, and surgery is the most effective treatment. Conventional open surgery is required to remove the posterior structures of the spine, which would lead to fracture of the posterior tension band, soft tissue injury, spine instability, and even spine deformity. So it is very important to protect and rebuild the posterior tension band for the stability of the spine. The team of Dr. John P. Kostuik from the Department of Orthopedics and Neurosurgery, the Johns Hopkins University, firstly introduced minimally invasive surgery for cervical and lumbar degenerative disease. However it has not been applied to the treatment of intra-spinal canal tumors. To date, the microsurgery of intra-spinal tumor through the trans-Quadrant channel pathway has not been widely performed in clinical practice. The investigators performed the microsurgery of intra-spinal canal tumor through the trans-Quadrant pathway in some patients previously and succeeded in the surgical treatments. The investigators analyzed the clinical data retrospectively, including surgical incision length, the volume of bleeding during operation, post-operative drainage volume, post-operative out-of-bed time point, post-operative length of stay in hospital, and post-operative visual analog pain (VAP) score. The group of patients using microsurgical technique through trans-Quadrant channel pathway showed better outcome compared with the group of patients using conventional open surgery. This innovation of microsurgery showed fewer traumas and bleeding, more rapid recovery, better prognosis and more safety in practice. Since there are some limitations to the retrospective study, it is necessary to design a prospective randomized controlled trial of the treatment of intra-spinal canal tumors using microsurgical technique through trans-Quadrant channel pathway.

DETAILED DESCRIPTION:
This study is the prospective randomized controlled clinical trial.

1. Patient Recruitment: Patients who meets the diagnostic criteria of intra-spinal canal tumor and has surgical indications from May 2016 to June 2018 in the department of neurosurgery of our hospital could be recruited.
2. Screening: Demographic characteristics, such as gender, age, history of diseases (including but not limited in diabetes, heart disease, smoking history, and operation history, etc.), related laboratory tests (blood routing test, liver and kidney functions, electrolytes, blood coagulation function, and ECG, etc.) before entering either group.
3. Grouping: Patients who meets the diagnostic criteria and does not meet the exclusion criteria would be assigned into the experimental group and control group randomly. The informed consent forms should be signed before grouping.
4. Surgery: Patients in the experimental group will receive operation using microsurgical techniques through trans-Quadrant channel pathway. Patients in the control group will receive conventional open surgery.
5. Post-operative Observation and Follow-up: Clinical data will be collected after surgery and during follow-up. The time points include the 1st day, 7th day, 30th day, 90th day, and 180th day after surgery.
6. Statistical Analysis: Statisticians are blinded to the clinical data and grouping. The software SPSS (V. 16.0) will be used in statistics.

ELIGIBILITY:
Inclusion Criteria:

* The patient should meet the diagnostic criteria of intra-spinal canal tumors and the indications for surgery. Meanwhile, the length of tumor should no more than 5 cm, and the cross-sectional area should be less than 2/3 of the respective area of the spinal canal.
* The patient was never be treated with any spinal surgery.
* There was no cognitive impairment before onset of diseases or other diseases which can cause cognitive dysfunction.
* The patient should sign the informed consent forms.

Exclusion Criteria:

* The patient is diagnozed as non intra-spinal canal tumors, spinal degenerative diseases, or other spinal diseases.
* The patient received spinal surgery previously.
* The patient suffered from serious heart, lung, liver, or kidney insufficiency.
* The patient has other spinal and spinal cord diseases rather than intra-spinal canal tumor, such as disc herniation, vertebral fractures.
* The patient has severe diabetes, coronary heart disease, coagulation disorders, difficult to correct before operation, or cannot tolerate surgery.
* The patient has other surgical contraindications.
* The patient is pregnant or breast-feeding.
* The patient is unable to sign the informed consent voluntarily.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Postoperational Length of Stay in Hospital | From the day after operation to up to 4 weeks after operation.
  The duration of hospital stay from the day after operation to the day of discharge.

SECONDARY OUTCOMES:
Operaion duration | On the day of operation.
  The time duration of operation.
Operative incision length | On the day of operation.
  The skin incision length of operation.
Blood loss in operation | On the day of the surgery.
  The blood lost during operatioin.
Cost of the surgery | On the day of the surgery.
  The cost of the surgery, including operation cost, blood cost, anesthetic cost, and material cost, etc.
Post-operative drainage volume | On the 1st day after operation.
  The drainage volume of surgery site from postoperation to the 1st day morning after operation.
Post-operative VAS | On the 7th day and 30th day after operation.
  The VAS scores on the 7th and 30th days after operation.
The improvement rate of Japanese Orthopaedic Association Scores (JOAS) | On the 1st day after operation.
  Collect the pre-operational JOAS score and the JOAS score on the 1st day after operation.
The improvement rate of JOAS | On the 7th day after operation.
  Collect the pre-operational JOAS score and the JOAS score on the 7th day after operation.
The improvement rate of JOAS | On the 30th day after operation.
  Collect the pre-operational JOAS score and the JOAS score on the 30th day after operation.
The improvement rate of JOAS | On the 90th day after operation.
  Collect the pre-operational JOAS score and the JOAS score on the 90th day after operation.
The improvement rate of JOAS | On the 180th day after operation.
  Collect the pre-operational JOAS score and the JOAS score on the 180th day after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Bao, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No